CLINICAL TRIAL: NCT06719505
Title: Comparison Between a Multicomponent Training Program and Pilates on Muscle Mass, Muscle Strength, and Physical Performance in Older Adults: A Randomized Controlled Trial
Brief Title: Multicomponent vs Pilates on Mass, Strength, and Physical Performance in Older Adults
Acronym: versus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do Norte do Parana (Other)
Responsible Party: Principal Investigator, Laís Campos de Oliveira, Doctor Teacher Laís Campos de Oliveira, Universidade Estadual do Norte do Parana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Multicomponent vs Pilates
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Muscle Mass; Muscle Strength; Physical Performance
Keywords: Aging; Elderly; Fragility; Physical exercise; Sarcopenia
MeSH Terms: conditions — Motor Activity; Sarcopenia

STUDY DESIGN:
Intervention Model Description: The interventions will last for six months, three times per week, for one hour, on non-consecutive days. The interventions for the Multicomponent group will consist of exercises for aerobic training, strengthening, resistance, balance, and flexibility, with one protocol for the first 3 months and a second protocol for months 4-6. The number of repetitions for each exercise will range from 3 sets of 8 to 10 repetitions, totaling 18 exercises. The Pilates exercise group will perform stretching and strengthening exercises targeting the main muscle groups, with one protocol for the first 3 months and a second protocol for months 4-6. Each protocol will consist of 17 exercises, with 3 sets of 8 to 10 repetitions.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The sample randomization will be conducted secretly by a professional who is unaware of the study and the volunteers. This professional will perform the randomization using random numbers to assign the study sample into two groups: the Multicomponent Group (EM) (n=50) and the Pilates Group (EP) (n=50). The same professional will then place the assignments in opaque envelopes, which will be sealed and contain the group allocation inside. Participants will be informed that they may be allocated to either group during the recruitment and selection process. Moreover, both the participants and the researchers will only know which group each individual is assigned to at the moment of envelope delivery.
  Assessments will be conducted before the intervention, during the treatment (3 months), and after its completion (6 months) by the same professional, who will be blinded to the identities of the volunteers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent exercises (ME) (Active Comparator): The interventions for the ME group will consist of exercises for aerobic training, strengthening, resistance, balance, and flexibility. The first week of the protocol will be dedicated to familiarizing the volunteers with the exercises, during which the correct execution of the movements will be demonstrated. Resources such as dumbbells, ankle weights, elastic bands, resistance bands, sticks, obstacles, and balls will be used.
  Interventions: Other: ME
- Pilates exercises (PE) (Experimental): For the intervention of the PE group, the first week of the protocol will be used to familiarize participants with the exercises, during which the correct execution of the movements will be demonstrated and each principle of the method will be explained: concentration, centering, precision, breathing, control, and fluidity. Regarding the progression of spring resistance, it will occur according to the volunteers' progress by switching to a spring with higher resistance (changing the position of the springs on the equipment or replacing them with ones of higher resistance). The basic equipment used will include the Cadillac Trapeze, Combo Chair, Universal Reformer, Ladder Barrel, and Wall Unit.
  Interventions: Other: PE

INTERVENTIONS:
Other: ME — Exercises selected with a focus on the major muscle groups. There will be one protocol for the first 3 months and a second protocol for months 4-6, with the number of repetitions for each exercise varying from 3 sets of 8 to 10 repetitions, totaling 18 exercises.
  Arms: Multicomponent exercises (ME)
Other: PE — The stretching and strengthening exercises will target the major muscle groups, and at the end of each session (lasting approximately 60 minutes), the instructor will guide the participant through a relaxation exercise using an EVA foam roller. The exercises were selected to improve overall muscle strength, as traditionally applied in Pilates. There will be one protocol for the first 3 months and a second protocol for months 4-6, with 17 exercises in each protocol, varying from 3 sets of 8 to 10 repetitions.
  Arms: Pilates exercises (PE)

SUMMARY:
Introduction: The aging process can result in several physiological changes, such as the loss of muscle mass, muscle strength, and physical performance, collectively defined as sarcopenia. Sarcopenia is considered one of the primary health challenges among older adults. To prevent this condition and improve related health outcomes, regular physical exercise is the most recommended strategy, with multicomponent exercises being particularly effective for older individuals. Pilates is another potential form of physical exercise that has gained popularity among older adults seeking to improve muscle mass, strength, and physical performance. However, significant gaps remain in the literature, with a notable lack of studies evaluating the efficacy of Pilates in improving sarcopenic outcomes. Objective: To compare the efficacy of multicomponent training programs versus Pilates in improving muscle mass, muscle strength, and physical performance in older adults. Methods: A total of 100 older adults aged 60 to 80 years, of both sexes, will be randomized into two intervention groups: the Multicomponent Training Group (n=50) and the Pilates Group (n=50). Evaluations will be conducted at three time points: baseline (before the intervention), mid-treatment (3 months), and post-treatment (6 months). The following instruments will be used: Dual-energy X-ray absorptiometry (DXA) will be used to assess muscle mass. Muscle strength will be evaluated using an isokinetic dynamometer for the lower limbs and a handgrip dynamometer for the upper limbs. Physical performance will be assessed through the Brazilian version of the Short Physical Performance Battery (SPPB), the gait speed test, and the Timed Up and Go (TUG) test. The Feeling Scale will be applied to determine the affective valence of the exercise programs. The Shapiro-Wilk test will be performed to check the normality of the data, Student's t-test or Mann-Whitney U test will be used depending on whether the distribution is parametric or non-parametric, and ANCOVA will be used to compare the groups post-intervention, considering a 95% confidence interval (p<0.05). The data will be analyzed using SPSS 25.0 software.

DETAILED DESCRIPTION:
The sample will consist of 100 elderly individuals of both sexes, aged between 60 and 80 years. The sample size calculation for this study was performed using the Bioestat 5.3 program, based on the values of whole-body DEXA (dual-energy X-ray absorptiometry) assessment, provided in a previous study (Seo et al., 2021). In this case, the post-intervention mean and standard deviation between the Resistance Training group (1566.75±189.47) and the Control group (maintaining routine habits) (1446.86 ± 206.42) were used, with a test power of 80%, an alpha value of 0.05, and a 15% error rate, which indicated the need for 50 participants in each group (Multicomponent Group and Pilates Group). Descriptive data analysis will be expressed as mean, standard deviation, and percentage delta of the difference. Normality will be assessed using the Shapiro-Wilk test. To verify if there are differences between the groups regarding baseline characteristics (age, weight, height, and BMI) at the pre-intervention stage, Student's t-test for independent samples or the Mann-Whitney U test will be used, depending on whether the data are parametric or non-parametric. To compare the groups post-intervention, ANCOVA will be used, with baseline data as covariates. If the data exhibit non-parametric characteristics, the Mann-Whitney U test will be applied to compare the groups based on the difference between pre- and post-intervention. A confidence interval of 95% (p<0.05) will be accepted. Data will be processed using SPSS 25.0 software. Effect sizes (Cohen's d) will be calculated and classified as small (0.20), medium (0.50), or large (0.80). For effect size calculations, the GPower 3.1 program will be used.

ELIGIBILITY:
Inclusion Criteria:

* Not currently participating in a physical training program for at least six months;
* No medical restrictions for physical activity and physical tests;
* Achieve a score of 19 or higher on the Mini-Mental State Examination.

Exclusion Criteria:

* Individuals with severe/disabling musculoskeletal and/or neurological dysfunctions;
* Neurological disorders or cognitive impairment;
* Use of supplements for muscle mass increase;
* History of recent fractures or surgeries and severe cardiorespiratory diseases.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
1. Dual-energy X-ray absorptiometry (DXA) | 6 months
  A high-precision reference standard used to measure lean muscle mass. The values will be calculated by the ratio of appendicular lean mass divided by the square of height in meters, with values lower than 7 kg/m² for men and 5.5 kg/m² for women confirming the diagnosis of low lean mass.
2. Biodex Isokinetic Dynamometer System | 6 months
  Evaluation of isokinetic muscle strength of the knee extensors and flexors. The assessment consists of knee extension and flexion (concentric/concentric) at an angular velocity of 60°/s, starting with the knee flexed at 90°. Three sets of five repetitions will be performed with a 30-second rest interval between sets, and the same procedure will be carried out with the left leg.
3. Hydraulic Hand Dynamometer | 6 months
  Evaluation of handgrip strength. The best value from three attempts will be used for each hand.
4. Brazilian Version of the Short Physical Performance Battery (SPPB) | 6 months
  A battery of tests to assess physical performance, including balance, gait speed, and chair rise tests. It has predictive validity and clinical applicability.
5. Gait Speed Test: Evaluation of gait speed through the 4-meter Walking Speed Test and the 6-Minute Walk Test (6MWT) | 6 months
  The 4-meter Walking Speed Test is used as a short-distance gait speed test, measuring habitual or maximum speed manually with a stopwatch or electronically with a device to measure the individual's walking time over a four-meter course. The 6MWT is a submaximal measure of aerobic capacity. Both tests are used to assess physical performance
6. Timed Up and Go (TUG) | 6 months
  A test used to assess physical function, commonly employed to evaluate the risk of falls. For the test, the time it takes for participants to rise from a chair, walk at a comfortable pace in a straight line for three meters, turn around, and return to the chair to sit down will be timed.

SECONDARY OUTCOMES:
7. Simple questionnaire to rapidly diagnose sarcopenia (SARC-F) | 6 months
  It is a validated and consistent questionnaire to identify people at risk of adverse outcomes due to sarcopenia. It consists of 5 items, self-reported by patients, based on the individual's perception of their strength limitations, ability to walk, get up from a chair, climb stairs and history of falls. Each item can be scored from 0 to 2, with 0 being no difficulty, 1 being some difficulty, and 2 being very difficult or unable to perform. In the falls item, 0 corresponds to no falls, 1 corresponds to 1 to 3 falls and 2 corresponds to 4 or more falls. The final score can range from 0 to 10, with a score of 4 being considered predictive of sarcopenia.
8. Mini Nutritional Assessment (MNA) | 6 months
  A screening tool for the nutritional status of participants, consisting of simple measures and six questions that can be answered in less than 5 minutes. It includes anthropometric measurements (body mass index, weight loss), global assessment (mobility), and dietary questionnaire and subjective evaluation (food intake, neuropsychological issues, acute illness). A score between 12-14 points indicates normal nutrition, 8-11 points indicates a risk of malnutrition, and 0-7 points indicates malnutrition.
9. Feeling Scale - Pleasure and Displeasure during Exercise | 6 months
  The affective valence scale will be used to measure participants' feelings of pleasure/affect related to the exercises. The score ranges from +5, indicating pleasure during exercise with a feeling of "very good," to -5, indicating displeasure with a feeling of "very bad" during exercise execution. The closer the score is to +5, the more pleasure the participant experiences while performing the exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Laís C. de Oliveira, PhD, Principal Investigator — UENP
Locations (1):
- Universidade, Jacarezinho, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bottaro M, Russo AF, de Oliveira RJ. The effects of rest interval on quadriceps torque during an isokinetic testing protocol in elderly. J Sports Sci Med. 2005 Sep 1;4(3):285-90. eCollection 2005 Sep 1. PMID 24453533
- [Background] Buckinx F, Aubertin-Leheudre M. Relevance to assess and preserve muscle strength in aging field. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Aug 30;94:109663. doi: 10.1016/j.pnpbp.2019.109663. Epub 2019 Jun 7. PMID 31176745
- [Background] Cruz-Jentoft AJ, Sayer AA. Sarcopenia. Lancet. 2019 Jun 29;393(10191):2636-2646. doi: 10.1016/S0140-6736(19)31138-9. Epub 2019 Jun 3. PMID 31171417
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Izquierdo M, Merchant RA, Morley JE, Anker SD, Aprahamian I, Arai H, Aubertin-Leheudre M, Bernabei R, Cadore EL, Cesari M, Chen LK, de Souto Barreto P, Duque G, Ferrucci L, Fielding RA, Garcia-Hermoso A, Gutierrez-Robledo LM, Harridge SDR, Kirk B, Kritchevsky S, Landi F, Lazarus N, Martin FC, Marzetti E, Pahor M, Ramirez-Velez R, Rodriguez-Manas L, Rolland Y, Ruiz JG, Theou O, Villareal DT, Waters DL, Won Won C, Woo J, Vellas B, Fiatarone Singh M. International Exercise Recommendations in Older Adults (ICFSR): Expert Consensus Guidelines. J Nutr Health Aging. 2021;25(7):824-853. doi: 10.1007/s12603-021-1665-8. PMID 34409961
- [Background] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony P, Charlton KE, Maggio M, Tsai AC, Grathwohl D, Vellas B, Sieber CC; MNA-International Group. Validation of the Mini Nutritional Assessment short-form (MNA-SF): a practical tool for identification of nutritional status. J Nutr Health Aging. 2009 Nov;13(9):782-8. doi: 10.1007/s12603-009-0214-7. PMID 19812868
- [Background] Mehmet H, Yang AWH, Robinson SR. Measurement of hand grip strength in the elderly: A scoping review with recommendations. J Bodyw Mov Ther. 2020 Jan;24(1):235-243. doi: 10.1016/j.jbmt.2019.05.029. Epub 2019 May 24. PMID 31987550
- [Background] Melo MO, Gomes LE, Silva YO, Bonezi A, Loss JF. Assessment of resistance torque and resultant muscular force during Pilates hip extension exercise and its implications to prescription and progression. Rev Bras Fisioter. 2011 Jan-Feb;15(1):23-30. PMID 21519714
- [Background] Oliveira LC, Pires-Oliveira DA, Abucarub AC, Oliveira LS, Oliveira RG. Pilates increases isokinetic muscular strength of the elbow flexor and extensor muscles of older women: A randomized controlled clinical trial. J Bodyw Mov Ther. 2017 Jan;21(1):2-10. doi: 10.1016/j.jbmt.2016.03.002. Epub 2016 Mar 10. PMID 28167180
- [Background] Seo MW, Jung SW, Kim SW, Lee JM, Jung HC, Song JK. Effects of 16 Weeks of Resistance Training on Muscle Quality and Muscle Growth Factors in Older Adult Women with Sarcopenia: A Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Jun 23;18(13):6762. doi: 10.3390/ijerph18136762. PMID 34201810
- See also: Approval of the Ethics Committee for Research with Human Beings in Brazil — http://plataformabrasil.saude.gov.br/login.jsf